CLINICAL TRIAL: NCT04935996
Title: A Study Pilot About the Contribution of Pleuropulmonary Echography Iin Acute Bronchiolitis Among Infants
Acronym: ECHOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/579
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pleuropulmonary echography (Experimental)
  Interventions: Device: Pleuropulmonary echography

INTERVENTIONS:
Device: Pleuropulmonary echography — Pleuropulmonary echography is performed, in addition of the chest X-ray already performed in routine care

SUMMARY:
Pleuropulmonary echography remains an almost non-existent tool in routine pediatric practice.

Our study is part of a desire to develop its use in pediatrics, in particular for the diagnosis of acute bacterial pneumonitis associated with acute bronchiolitis among infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged <= 2 years old
* Medical diagnosis of acute bronchiolitis requiring hospitalization in the pediatric departments of the Besançon University Hospital
* No opposition from the parents for performing the pleuropulmonary echography.

Exclusion Criteria:

* Children aged > 2 years old
* Infants aged < 2 years old consultant in pediatric emergencies for acute bronchiolitis without subsequent hospitalization.
* Previous chronic lung disease (including pulmonary bronchodysplasia), unoperated congenital heart disease or neuromuscular disease.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Comparison between PleuroPulmonary Echography [PPE] and pulmonary radiography | Day 1
  Comparative analysis between PPE and chest/pulmonary radiography (gold standard) for the diagnosis of bacterial pneumonitis associated with acute bronchiolitis in infants.

CONTACTS AND LOCATIONS:
Overall Officials: Julien BEHR, MD, Principal Investigator — CHU de Besançon

IPD SHARING:
Plan to Share IPD: No